CLINICAL TRIAL: NCT01760759
Title: Antiretroviral Therapy Adherence and Secondary Prevention of Human Immunodeficiency Virus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Carla Rash, Assistant Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-205O-2; R01HD075630 (NIH)
Record Dates: First submitted 2012-08-21; First posted 2013-01-04 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: HIV
Keywords: HIV; Antiretroviral therapy adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): Patients receive usual care from their medical providers.
- Usual care plus cell phone reminders (Experimental): Patients receive reminders, scheduled to occur daily at time(s) of scheduled antiretroviral therapy dosing.
  Interventions: Behavioral: cell phone reminders
- Usual care, reminders & contingency management for adherence (Experimental): Patients receive reminders and reinforcement in the form of vouchers for each video that they send in indicating adherence at the appropriate time.
  Interventions: Behavioral: cell phone reminders; Behavioral: contingency management for adherence

INTERVENTIONS:
Behavioral: cell phone reminders — Patients receive reminders, scheduled to occur daily at time(s) of scheduled antiretroviral therapy dosing.
  Arms: Usual care plus cell phone reminders; Usual care, reminders & contingency management for adherence
Behavioral: contingency management for adherence — Patients will receive reinforcement in the form of vouchers for each video that they send in indicating adherence at the appropriate time.
  Arms: Usual care, reminders & contingency management for adherence

SUMMARY:
In this study, investigators propose to randomize 165 human immunodeficiency virus positive patients to one of three 16-week treatment conditions: (1) standard care; (2) standard care + cell phone-based adherence reminders; or (3) standard care + cell phone-based adherence reminders and contingency management. In this latter condition, patients will earn reinforcement for sending in time- and date-stamped self videos of antiretroviral therapy medication ingestion. Primary outcomes will include viral loads and self-report measures of adherence, and effects will be evaluated both during the treatment period and throughout a one-year follow-up. Investigators hypothesize that the cell phone reminder condition will improve adherence relative to standard care, and the cell phone reminder plus contingency management condition will have the best outcomes. Results from this study may have widespread implications for the use of cell phones as a novel technology to improve initial adherence to antiretroviral therapy, thereby reducing the spread of drug resistant human immunodeficiency virus strains to the community.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* initiating or on an antiretroviral therapy regimen and have a viral load >200 copies/mL in the past 6 months
* one or more risk factors for poor adherence
* English speaking
* willing to use a cell phone to receive reminders and record medication ingestion for up to 16 weeks
* able to read at 5th grade level and pass a brief quiz related to understanding the informed consent form

Exclusion Criteria:

* living in an environment or has a visiting nurse that dispenses antiretroviral therapy medication
* participating in another antiretroviral therapy adherence study
* uncontrolled psychiatric disorders
* significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
change in copies of human immunodeficiency virus per milliliter | Week 48
self-report of medication adherence | baseline
self-report of medication adherence | Week 8
self-report of medication adherence | Week 16
self-report of medication adherence | Week 24
self-report of medication adherence | Week 36
self-report of medication adherence | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Carla Rash, Ph.D., Principal Investigator — UConn Health
Locations (2):
- United States (2):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Nathan Smith Clinic, Yale-New Haven Hospital, New Haven, Connecticut